CLINICAL TRIAL: NCT01765998
Title: The Effect of Probiotics on the Rate of Recovery of Inflammatory Bowel Disease Exacerbation (Crohn's Disease) and Markers of Inflammation
Brief Title: The Effect of Probiotics on Exacerbation of Inflammatory Bowel Disease Exacerbation (Crohn's Disease)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Arnon Blum, Doctor, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18-2012.CTIL
Record Dates: First submitted 2013-01-06; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, endothelial progenitor cells, probiotic
MeSH Terms: conditions — Crohn Disease | interventions — Probiotics; Powders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): To study the effect of probiotic on the ability to build endothelial progenitor stem cells and to study clinical recovery of patients with Crohn's Disease.
  Interventions: Drug: Probiotic
- placebo (Placebo Comparator): This will be the comparison group to the experimantal group that recives Probiotic.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic — Clinical evaluation according to the Crohn's activity scale
  Other Names: Bio 25; powder in HPMC Capsule
  Arms: Probiotic
Drug: Placebo
  Arms: placebo

SUMMARY:
Inflammatory Bowel Disease (IBD) is an immune mediated chronic intestinal condition. It includes ulcerative colitis (UC) and Crohn's disease(CD). probiotics have been shown to be effective in varried clinical conditions ranging fron infantile diarrhea, necrotizing enterocolitis,helicobacter pylori infections, etc.

DETAILED DESCRIPTION:
This is a prospective study that will enroll 50 patients with Crohn's disease.Each patient will get the study medication for 6 weeks and will be evaluated twice- before enrollment and after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohns' disease who are stable or have mild acute exacerbations that do not necessitate treatment with systemic corticosteroids

Exclusion Criteria:

* pregnant women, under 18 years or over 60 years,
* patients with known ulcerative colitis,
* patients with any cancer,
* patients with heart failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
endothelial stem cells | one year
  to study the ability to create endothelial progenitor stem cells following probiotic management compared to placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Blum, MD, Principal Investigator — Baruch Padeh Medical Center
Locations (1):
- Baruch Padeh Medical Center, Tiberias, Lower Galilee, Israel